CLINICAL TRIAL: NCT00525837
Title: Systematic Assessment of Response to Open-label Treatment With Varenicline in Depressed Outpatient Smokers
Brief Title: Study of Mood Effects of Varenicline (Chantix) in Depressed Outpatient Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: Brown University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0707-002
Record Dates: First submitted 2007-09-04; First posted 2007-09-06 (Estimated); Results first posted 2011-05-23 (Estimated); Last update posted 2018-11-28 (Actual); Status verified 2018-10

CONDITIONS: Depressive Disorder; Smoking
Keywords: varenicline; depression; anhedonia; smoking
MeSH Terms: conditions — Depressive Disorder; Smoking; Depression; Anhedonia | interventions — Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- varenicline (Other): open label varenicline
  Interventions: Drug: fixed dose varenicline; Drug: varenicline

INTERVENTIONS:
Drug: fixed dose varenicline — varenicline 0.5 mg po daily for days 1-3, 0.5 twice daily for days 4-7, 1 mg twice daily thereafter for study duration.
  Other Names: Chantix
Drug: varenicline — up to 1 mg twice daily
  Other Names: Chantix

SUMMARY:
This study will assess whether varenicline (chantix) has antidepressant properties when used in addition to other psychiatric medication. It will also assess whether varenicline improves the inability to feel pleasure (i.e. anhedonia), and if it is well-tolerated when used with psychiatric medications.

Enrolled patients will be assessed for improved mood, improved anhedonia, overall sense of health, side effects as well as tobacco use for 6-8 weeks.

Medication will be provided free of charge.

DETAILED DESCRIPTION:
Outpatient smokers who are depressed despite current stable psychiatric medication regimens will be invited to participate.

They will receive varenicline dosed according to FDA-approved smoking cessation regime; patients will be assessed using QIDS-SR16, snaith-hamilton anhedonia rating scale, SAFTEE and clinical global improvement self-report scales and clinician global improvement scales at the above time intervals.

Concurrent medication, psychiatric and non-psychiatric, will be recorded, as will vital signs (BP, HR, weight) and tobacco use.

ELIGIBILITY:
Inclusion Criteria:

1. Meets DSM-IV symptoms criteria for a mood disorder including major depression [unipolar or bipolar], depressive disorder NOS, dysthymia, adjustment disorder with depressed mood, or substance-induced mood disorder.
2. Failed to achieve full symptom remission with previous pharmacotherapy.
3. Current tobacco users.
4. Able to give written, informed consent.

Exclusion Criteria:

1. Past adverse reaction to varenicline.
2. Renal failure or dialysis.
3. Current pregnancy or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-09; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noah S Philip, MD, Principal Investigator — Butler Hospital; Lawrence H Price, MD, Study Director — Butler Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Philip NS, Carpenter LL, Tyrka AR, Whiteley LB, Price LH. Varenicline augmentation in depressed smokers: an 8-week, open-label study. J Clin Psychiatry. 2009 Jul;70(7):1026-31. doi: 10.4088/jcp.08m04441. Epub 2009 Mar 24. PMID 19323966

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Varenicline
Started | 18
Completed | 14
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Varenicline
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (10.1)
Age, Customized [Number; unit: participants]
  Between 18 and 65 years | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Quick Inventory of Depressive Symptoms, 16 Question Self-report
Description: this is a 16-item self report questionnaire that measures depressive symptoms.
  Improvement is reported in change in depressive score
  score ranges from 0-27, with higher numbers indicating more severe symptom reporting.
  change is calculated by baseline plus/minus the value at the later time point
Time Frame: Baseline and every 2 weeks until 8 weeks or study endpoint
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Varenicline
Number analyzed (Participants) | 18
Units on a scale | 4.7 [2.6 to 6.8]

2. Secondary Outcome: Improvement on Snaith-Hamilton Pleasure Scale (SHAPS)
Description: Snaith-Hamilton Pleasure Scale (SHAPS; Snaith et al, 1995). The SHAPS is a 14-item scale that measures anhedonia, the inability to experience pleasure. The items cover the domains of: social interaction, food and drink, sensory experience, and interest/pastimes. A score of 2 or less constitutes a "normal" score, while an "abnormal" score is defined as 3 or more. Each item has four possible responses: strongly disagree, disagree, agree, or strongly agree. Either of the "disagree" responses score one point, and either of the "agree" responses score 0 points. Thus, the final score ranges from 0 to 14. The SHAPS has adequate construct validity and satisfactory test-retest reliability (ICC=0.70) (Franken et al, 2007). High internal consistency has also been reported (Cronbach's alpha of 0.94) (Franken et al, 2007)
Time Frame: 6-8 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Varenicline
Number analyzed (Participants) | 18
score on a scale | 24.9 (7.4)

3. Secondary Outcome: Improvement on Patient and Clinician Clinical Global Impression Rating Scale (CGI)
Description: Reference:
  Guy W, editor. ECDEU Assessment Manual for Psychopharmacology. 1976. Rockville, MD, U.S. Department of Health, Education, and Welfare
  The CGI is rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through to 7 (amongst the most severely ill patients).
Time Frame: 6-8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Varenicline
Number analyzed (Participants) | 14
units on a scale | 2.1 (1.4)

ADVERSE EVENTS:
Arm/Group | Varenicline
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 4/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=18)
gastrointestinal distress (Gastrointestinal disorders) | 3 (3)
insomnia (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No